CLINICAL TRIAL: NCT02401048
Title: A Multi-Center Open-Label Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib, in Combination With MEDI4736, in Subjects With Relapsed or Refractory Lymphomas
Brief Title: A Multi-Center Study of Ibrutinib in Combination With MEDI4736 in Subjects With Relapsed or Refractory Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: AstraZeneca (Industry); Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1136-CA
Record Dates: First submitted 2015-03-04; First posted 2015-03-27 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Diffuse Large B-Cell Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — ibrutinib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1b/ 2: Follicular lymphoma expansion cohort (Experimental): In the Phase 1b (safety portion) of the study, a starting dose of 560 mg of ibrutinib and 10 mg/kg of MEDI4736 explored in cohort 1 and followed a 6+3 dose de-escalation design. Phase 2 used the phase 1b starting dose.
  Interventions: Drug: Ibrutinib; Drug: MEDI4736
- Phase 1b/ 2: Diffuse large B-cell lymphoma expansion cohort (Experimental): In the Phase 1b (safety portion) of the study, a starting dose of 560 mg of ibrutinib and 10 mg/kg of MEDI4736 explored in cohort 1 and followed a 6+3 dose de-escalation design. Phase 2 used the phase 1b starting dose.
  Interventions: Drug: Ibrutinib; Drug: MEDI4736

INTERVENTIONS:
Drug: Ibrutinib
Drug: MEDI4736

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of the combination treatment of ibrutinib and MEDI4736 in subjects with relapsed or refractory lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented relapsed or refractory diffuse large B-cell lymphoma (DLBCL) or follicular lymphoma (FL)
* Measurable disease sites on CT scan (>1.5 cm in longest dimension)
* Adequate hematologic function:

  1. Absolute Neutrophil Count >1500 cells/mm3
  2. Platelets >50000 cells/mm3
  3. Hemoglobin >8.0 g/dL
* Adequate hepatic and renal function:

  1. AST or ALT ≤2.5 x ULN
  2. Bilirubin ≤1.5 x ULN
  3. Estimated creatinine clearance (Cockcroft-Gault) >40 mL/min
* ECOG 0 or 1

Exclusion Criteria:

* Received prior therapies: ibrutinib, or other BTK inhibitor and/or anti-PD1, anti-PD-L1, anti-PD-L2, anti-CD137, or CTLA-4 antibody
* Requires treatment or prophylaxis with a strong cytochrome P450 (CYP) 3A inhibitor
* Primary CNS lymphoma or evidence of CNS involvement by lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-05; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Liu, Study Director — Pharmacyclics LLC.
Locations (11):
- United States (11):
  - Site-0397, Birmingham, Alabama
  - Site-0047, Duarte, California
  - Site-0038, Stanford, California
  - Site-0388, Miami, Florida
  - Site-0126, Chicago, Illinois
  - Site-0020/0173, Boston, Massachusetts
  - Site-0729, Ann Arbor, Michigan
  - Site-0130, Detroit, Michigan
  - Site-0343, Hackensack, New Jersey
  - Site-0402, Philadelphia, Pennsylvania
  - Site-0114, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While the study include Phase 1b and 2, the dosing was not changed between phases (following the study design because there were no DLTs and thus no dose adjustments in from Phase 1b to Phase 2). Thus the study data were reported with Phases 1b and 2 combined.
Period: Overall Study
Arm/Group | Phase 1b/ 2: Follicular Lymphoma Expansion Cohort | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort
Started | 27 | 34
Completed | 5 | 4
Not Completed | 22 | 30

BASELINE CHARACTERISTICS:
Groups:
- Phase 1b/2: Follicular Lymphoma Expansion Cohort:; Phase 1b/2: Diffuse Large B-cell Lymphoma Expansion Cohort:: All participants who received at least one dose of study treatment.
- Total: Total of all reporting groups
Arm/Group | Phase 1b/2: Follicular Lymphoma Expansion Cohort: | Phase 1b/2: Diffuse Large B-cell Lymphoma Expansion Cohort: | Total
Number analyzed (Participants) | 27 | 34 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 15 | 34
  >=65 years | 8 | 19 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11.88) | 61.2 (15.15) | 59.3 (13.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 17 | 21 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 23 | 32 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 27 | 34 | 61

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b/2 : Overall Response Rate of Number of Participants
Description: The response criteria is measured based on the revised criteria for malignant lymphoma described by the International Working Group for NHL (Cheson 2014).
Time Frame: From the date of first study treatment until progressive disease
Population: While the study include Phase 1b and 2, the dosing was not changed between phases (following the study design because there were no DLTs and thus no dose adjustments in from Phase 1b to Phase 2). Thus the study data were reported with Phases 1b and 2 combined.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b/ 2: Follicular Lymphoma Expansion Cohort; Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort: All participants who received at least one dose of study treatment.
Arm/Group | Phase 1b/ 2: Follicular Lymphoma Expansion Cohort | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort
Number analyzed (Participants) | 27 | 34
Participants | 7 | 8

2. Secondary Outcome: Phase 1b/ 2: Duration of Response
Time Frame: Time from the date of initial response to the date of disease progression or the date of death due to any cause, whichever occurs first.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b/ 2: Follicular Lymphoma Expansion Cohort | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort
Number analyzed (Participants) | 7 | 8
Months | 11.3 [8.3 to NA] — The 95% Confidence Interval is not applicable because the median Duration of Response was estimated based on time to event data. The 95% Confidence limit cannot be estimated. | NA [2.5 to NA] — The median Duration of Response was not reached. The 95% Confidence limit cannot be estimated.

3. Secondary Outcome: Phase 1b/ 2: Progression-free Survival (PFS)
Time Frame: first dose date of study drug (ibrutinib or MEDI4736) to the first documentation of disease progression
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b/ 2: Follicular Lymphoma Expansion Cohort | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort
Number analyzed (Participants) | 27 | 34
Months | 10.2 [4.7 to 13.1] | 2.6 [1.5 to 4.4]

4. Secondary Outcome: Phase 1b/2: Overall Survival
Time Frame: First dose date of study drug (ibrutinib or MEDI4736) to the date of death due to any cause
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b/ 2: Follicular Lymphoma Expansion Cohort | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort
Number analyzed (Participants) | 27 | 34
Months | NA [23.6 to NA] — The median Overall Survival was not reached. The 95% Confidence limit cannot be estimated. | 5.1 [3.7 to 10.1]

5. Secondary Outcome: Phamacokinetics: Mean Maximum Observed Plasma Concentration (Cmax) for Ibrutinib
Description: Maximum observed plasma concentration of ibrutinib during the dosing interval on Lead-In Day 6/7 (ibrutinib only) or Cycle 3 Day 1 (ibrutinib + MEDI)
Time Frame: Lead-In Day 6/7 or Cycle 3 Day 1 (collected at predose, 1, 2, 4, and 6 hours post-dose)
Population: All subjects who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Phase 1b/ 2: Follicular Lymphoma Expansion Cohort; Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort: All participants who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Arm/Group | Phase 1b/ 2: Follicular Lymphoma Expansion Cohort | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort
Number analyzed (Participants) | 27 | 28
ng/mL
  Lead-In Day 6/7 | 196 (245) | 140 (117)
  Cycle 3 Day 1: number analyzed (Participants) | 19 | 7
  Cycle 3 Day 1 | 155 (102) | 183 (101)

6. Secondary Outcome: Pharmacokinetics: Mean Time to Maximum Observed Plasma Concentration (Tmax) for Ibrutinib
Description: Time to corresponding maximum observed plasma concentration of ibrutinib during the dosing interval on Lead-In Day 6/7 (ibrutinib only) or Cycle 3 Day 1 (ibrutinib + MEDI)
Time Frame: Lead-In Day 6/7 or Cycle 3 Day 1 (collected at predose, 1, 2, 4, and 6 hours post-dose)
Population: All subjects who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b/ 2: Follicular Lymphoma Expansion Cohort | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort
Number analyzed (Participants) | 27 | 28
hour
  Lead-In Day 6/7 | 1.95 [0.750 to 4.00] | 2.01 [0.930 to 6.00]
  Cycle 3 Day 1: number analyzed (Participants) | 19 | 7
  Cycle 3 Day 1 | 2.00 [1.00 to 6.05] | 2.07 [1.00 to 4.97]

7. Secondary Outcome: Pharmacokinetics: Mean Area Under the Plasma Concentration-Time Curve From Time 0-24 Hours (AUC0-24h) for Ibrutinib
Description: Ibrutinib AUC0-24h calculated using linear trapezoidal summation after dosing from time 0 to 24 hours on Lead-In Day 6/7 (ibrutinib only) or Cycle 3 Day 1 (ibrutinib + MEDI)
Time Frame: Lead-In Day 6/7 or Cycle 3 Day 1 (collected at predose, 1, 2, 4, and 6 hours post-dose)
Population: All subjects who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Phase 1b/ 2: Follicular Lymphoma Expansion Cohort | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort
Number analyzed (Participants) | 27 | 28
ng*h/mL
  Lead-In Day 6/7: number analyzed (Participants) | 26 | 27
  Lead-In Day 6/7 | 1078 (1013) | 936 (691)
  Cycle 3 Day 1: number analyzed (Participants) | 16 | 7
  Cycle 3 Day 1 | 1096 (748) | 1606 (901)

8. Secondary Outcome: Pharmacokinetics: Mean Terminal Elimination Half-Life (t1/2,Term) for Ibrutinib
Description: Ibrutinib terminal elimination half-life associated with the terminal slope (λz) of the semi-logarithmic plasma concentration-time curve, calculated as 0.693/λz on Lead-In Day 6/7 (ibrutinib only) or Cycle 3 Day 1 (ibrutinib + MEDI)
Time Frame: Lead-In Day 6/7 or Cycle 3 Day 1 (collected at predose, 1, 2, 4, and 6 hours post-dose)
Population: All subjects who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Phase 1b/ 2: Follicular Lymphoma Expansion Cohort | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort
Number analyzed (Participants) | 27 | 28
hour
  Lead-In Day 6/7: number analyzed (Participants) | 15 | 15
  Lead-In Day 6/7 | 5.35 (2.16) | 6.43 (1.92)
  Cycle 3 Day 1: number analyzed (Participants) | 7 | 3
  Cycle 3 Day 1 | 6.14 (1.96) | 5.27 (1.21)

9. Secondary Outcome: Pharmacokinetics: Mean Peak Plasma Concentration (Cmax) for MEDI4736
Description: Peak plasma concentration of MEDI4736 on Cycle 6 Day 1 (ibrutinib + MEDI)
Time Frame: Cycle 6 Day 1 (collected 10 minutes after end of infusion)
Population: All subjects who received at least one dose of study treatment and had evaluable pharmacokinetic data. Result data for both cohorts was pre-specified to be combined, and was not reported separately.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- Phase 1b/ 2: Follicular Lymphoma & DLBCL Expansion Cohort: All participants who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Arm/Group | Phase 1b/ 2: Follicular Lymphoma & DLBCL Expansion Cohort
Number analyzed (Participants) | 17
ug/mL | 388 (14.1)

10. Secondary Outcome: Pharmacokinetics: Mean Trough Plasma Concentration (Ctrough) for MEDI4736
Description: Trough plasma concentration of MEDI4736 on Cycle 6 Day 1 (ibrutinib + MEDI)
Time Frame: Cycle 6 Day 1 (predose)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Phase 1b/ 2: Follicular Lymphoma & DLBCL Expansion Cohort
Number analyzed (Participants) | 20
ug/mL | 207 (12.8)

11. Secondary Outcome: Pharmacokinetics: MEDI4736 Accumulation Ratio for Cmax
Description: Accumulation ratio from Cycle 6 Day 1 to Cycle 1 Day 1 for Cmax for MEDI4736
Time Frame: Cycle 6 Day 1 (collected 10 minutes after end of infusion)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Phase 1b/ 2: Follicular Lymphoma & DLBCL Expansion Cohort
Number analyzed (Participants) | 17
ratio | 1.90 (0.51)

12. Secondary Outcome: Pharmacokinetics: MEDI4736 Accumulation Ratio for Ctrough
Description: Accumulation ratio from Cycle 6 Day 1 to Cycle 1 Day 1 for Ctrough for MEDI4736
Time Frame: Cycle 6 Day 1 (predose)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Phase 1b/ 2: Follicular Lymphoma & DLBCL Expansion Cohort
Number analyzed (Participants) | 19
ratio | 3.31 (0.8)

13. Secondary Outcome: Bruton Tyrosine Kinase (BTK) Occupancy
Description: BTK occupancy
Time Frame: ibrutinib Lead-in Day 6 or 7 pre-dose
Population: All participants who received at least one dose of study treatment and had evaluable pharmacodynamics data.
Measure: Mean (Standard Error); unit: BTK % occupancy
Groups:
- Phase 1b/ 2: Follicular Lymphoma Expansion Cohort; Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort: All participants who received at least one dose of study treatment and had evaluable pharmacodynamics data.
Arm/Group | Phase 1b/ 2: Follicular Lymphoma Expansion Cohort | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort
Number analyzed (Participants) | 18 | 22
BTK % occupancy | 77.6 (8.4) | 91.2 (3.4)

14. Secondary Outcome: Pharmacodynamics of Ibrutinib in Subjects With Relapsed or Refractory Lymphomas
Description: BTK occupancy
Time Frame: Cycle 3 Day 1 Pre-dose
Population: All participants who received at least one dose of study treatment and had evaluable pharmacodynamics data.
Measure: Mean (Standard Error); unit: BTK % occupancy
Arm/Group | Phase 1b/ 2: Follicular Lymphoma Expansion Cohort | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort
Number analyzed (Participants) | 14 | 6
BTK % occupancy | 83.1 (9.4) | 94.4 (3.1)

15. Secondary Outcome: Pharmacodynamics of MEDI4736 in Subjects With Relapsed or Refractory Lymphomas
Description: Detectable Free Serum PD-L1 level
Time Frame: Cycle 3 Day1 Pre-dose
Population: In Follicular lymphoma expansion cohort, 7 subjects are below limit of quantitation. In Diffuse large B-cell lymphoma expansion cohort, all subjects below limit of quantitation.
Measure: Number; unit: pg/mL
Arm/Group | Phase 1b/ 2: Follicular Lymphoma Expansion Cohort | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort
Number analyzed (Participants) | 8 | 6
pg/mL | 18.4 | NA — NA means the data is not evaluable

ADVERSE EVENTS:
Time Frame: All AEs, whether serious or non-serious, are documented in the source documents from the time the signed and dated ICF is obtained until 30 days following the last dose of ibrutinib and 90 days following the last dose of MEDI4736.
Groups:
- Phase 1b/2: Follicular Lymphoma Expansion Cohort:; Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort:: All subjects who received at least one dose of study treatment.
Arm/Group | Phase 1b/2: Follicular Lymphoma Expansion Cohort: | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort:
All-Cause Mortality (participants affected / at risk) | 6/27 | 24/34
Serious Adverse Events (participants affected / at risk) | 10/27 | 23/34
Other Adverse Events (participants affected / at risk) | 27/27 | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b/2: Follicular Lymphoma Expansion Cohort: (N=27) | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort: (N=34)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (3) | 3 (4)
Left Ventricular Failure (Cardiac disorders) | 0 (0) | 1 (1)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 6 (7)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b/2: Follicular Lymphoma Expansion Cohort: (N=27) | Phase 1b/ 2: Diffuse Large B-cell Lymphoma Expansion Cohort: (N=34)
Neutropenia (Blood and lymphatic system disorders) | 6 (13) | 11 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 6 (11)
Increased tendancy to bruise (Blood and lymphatic system disorders) | 5 (7) | 4 (5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 6 (8)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (7)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 3 (3)
Dry eye (Eye disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 16 (23) | 16 (27)
Nausea (Gastrointestinal disorders) | 9 (9) | 12 (15)
Constipation (Gastrointestinal disorders) | 3 (3) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 4 (5) | 6 (6)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 6 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 4 (5) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 4 (5)
Fatigue (General disorders) | 12 (13) | 16 (19)
Oedema peripheral (General disorders) | 7 (10) | 13 (22)
Pyrexia (General disorders) | 3 (3) | 6 (7)
Peripheral swelling (General disorders) | 2 (2) | 2 (4)
Upper respiratory tract infection (Infections and infestations) | 12 (19) | 3 (4)
Urinary tract infection (Infections and infestations) | 3 (5) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 3 (6)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 4 (6)
Blood creatinine increased (Investigations) | 1 (2) | 3 (9)
Weight decreased (Investigations) | 2 (2) | 2 (3)
Weight increased (Investigations) | 0 (0) | 4 (7)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 11 (11)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (6) | 5 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (4) | 5 (8)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (6) | 4 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (9) | 5 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (9) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (8)
Dizziness (Nervous system disorders) | 3 (4) | 6 (7)
Headache (Nervous system disorders) | 6 (10) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 4 (7) | 2 (2)
Dysguesia (Nervous system disorders) | 2 (2) | 3 (3)
Memory impairment (Nervous system disorders) | 3 (3) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (4) | 3 (3)
Somnolence (Nervous system disorders) | 3 (4) | 1 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 6 (7)
Anxiety (Psychiatric disorders) | 5 (5) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 6 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (14) | 7 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4)
Oropharyngeal (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (13) | 7 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (7)
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 2 (6) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-02-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT02401048/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT02401048/SAP_001.pdf